CLINICAL TRIAL: NCT04968873
Title: Common Bile Duct Pressure After Intraoperative Instrumentation in Patients With Uncomplicated Choledocholithiasis
Brief Title: Common Bile Duct Pressure After Surgical Exploration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos R. Cervantes Sanchez (Other Government)
Responsible Party: Sponsor-Investigator, Carlos R. Cervantes Sanchez, General Surgery Service, Hospital General de Chihuahua - Dr. Salvador Zubirán Anchondo
Organization: Hospital General de Chihuahua - Dr. Salvador Zubirán Anchondo (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2001/0023
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Choledocholithiasis
Keywords: Choledocholithiasis; common bile duct; cholangiogram.
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Choledocholithiasis (Experimental): Patients were managed by elective open cholecystectomy and operative exploration of the common bile duct.
  Interventions: Procedure: Cholecystectomy and common bile duct exploration

INTERVENTIONS:
Procedure: Cholecystectomy and common bile duct exploration — During elective open cholecystectomy, a basal commcn dile duct (CBD) manometry was obtained immediately after cholecystectomy, with a 10 Fr. silicone T tube introduced into the cystic duct and connected to a glass manometer.

SUMMARY:
A study that included patients of any gender between 15 and 70 years, with the diagnosis of choledocholithiasis who required a cholecystectomy with an exploration of bile ducts. Conventional cholecystectomy was performed and a T-tube was inserted in the common bile duct (CBD) to measure the intraluminal pressure immediately after the procedure, and weekly thereafter, with a 6-week follow-up. A control T-tube radiological study was performed at six weeks to exclude residual stones.

DETAILED DESCRIPTION:
A clinical, controlled, prospective, longitudinal, descriptive, observational and double-blinded study was designed. Patients of any gender between 15 and 70 years, with a diagnosis of choledocholithiasis, and who required a cholecystectomy with an exploration of bile ducts were included. Conventional cholecystectomy was performed and perioperative T-tube CBD pressure was registered immediately after the procedure, and weekly thereafter, with a 6-week follow-up.

Control T-tube cholangiogram was performed at six weeks to exclude residual stones. Data was analyzed with T-test for parametric values.

ELIGIBILITY:
Inclusion Criteria: Choledocholithiasis -

Exclusion Criteria: To not complete the follow-up period

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-03 (Actual); Primary Completion 2001-08 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Basal common bile duct (CBD) pressure | Intraoperative
  Basal CBD manometry was obtained immediately after cholecystectomy
First week control common bile duct pressure | First week
  CBD manometry was obtained one week after cholecystectomy
Second week control common bile duct pressure | Second week
  CBD manometry was obtained two weeks after cholecystectomy
Third week control common bile duct pressure | Third week
  CBD manometry was obtained three weeks after cholecystectomy
Fourth week control common bile duct pressure | Fourth week
  CBD manometry was obtained four weeks after cholecystectomy
Fifth week control common bile duct pressure | Fifth week
  CBD manometry was obtained five weeks after cholecystectomy
Sixth week control common bile duct pressure | Sixth week
  CBD manometry was obtained six weeks after cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: David Saldaña-Cortés, MD, Principal Investigator — General Surgery Service

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When summary data are published
Access Criteria: All information should be requested from the corresponding author.

REFERENCES:
- [Background] Mendez-Sanchez N, Jessurun J, Ponciano-Rodriguez G, Alonso-de-Ruiz P, Uribe M, Hernandez-Avila M. Prevalence of gallstone disease in Mexico. A necropsy study. Dig Dis Sci. 1993 Apr;38(4):680-3. doi: 10.1007/BF01316800. PMID 8462367
- [Background] González-Pérez LG, Zaldívar-Ramírez FR, Tapia-Contla BR, Díaz-Contreras-Piedras CM, Arellano-López PR, Hurtado-López LM. Factores de riesgo de la coledocolitiasis asintomática; experiencia en el Hospital General de México. Cir Gen. 2018;40(3):164-168.
- [Background] Csendes A, Sepulveda A, Burdiles P, Braghetto I, Bastias J, Schutte H, Diaz JC, Yarmuch J, Maluenda F. Common bile duct pressure in patients with common bile duct stones with or without acute suppurative cholangitis. Arch Surg. 1988 Jun;123(6):697-9. doi: 10.1001/archsurg.1988.01400300039005. PMID 3369934
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Csendes A, Kruse A, Funch-Jensen P, Oster MJ, Ornsholt J, Amdrup E. Pressure measurements in the biliary and pancreatic duct systems in controls and in patients with gallstones, previous cholecystectomy, or common bile duct stones. Gastroenterology. 1979 Dec;77(6):1203-10. No abstract available. PMID 499707
- [Result] Copelan A, Kapoor BS. Choledocholithiasis: Diagnosis and Management. Tech Vasc Interv Radiol. 2015 Dec;18(4):244-55. doi: 10.1053/j.tvir.2015.07.008. Epub 2015 Jul 15. PMID 26615165